CLINICAL TRIAL: NCT01492530
Title: Reducing HIV Risk Behaviors and Psychosocial Stressors Among Bisexual African American Men
Brief Title: Men of African American Legacy Empowering Self
Acronym: MAALES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); California HIV/AIDS Research Program (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nina Harawa, Associate Professor, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AL04-DREW-840; 2P20MD000182 (NIH)
Record Dates: First submitted 2011-12-09; First posted 2011-12-15 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: HIV
Keywords: Men who have sex with Men and Women; HIV Prevention; Behavioral Intervention; Condom use; African American MSMW
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6-session, small group (Experimental): Men of African American Legacy Empowering Self (MAALES) Intervention, a six-session, theoretically grounded, small-group intervention held over 3 weeks. Includes an additional 2 booster sessions at 6 and 18 weeks following Session 6.
  Interventions: Behavioral: Men of African American Legacy Empowering Self
- HIV Education & Risk Reduction Session (Active Comparator): 20-30 minute standard, client-centered HIV education and risk-reduction session administered over the phone or in person. Similar to that received during pre-test counseling for HIV testing.
  Interventions: Behavioral: Standard HIV Education & Risk Reduction

INTERVENTIONS:
Behavioral: Men of African American Legacy Empowering Self — Small group intervention. 6 main sessions + 2 booster sessions. Each session lasts 2 hours. Main sessions held over 3 weeks.
  Other Names: MAALES
  Arms: 6-session, small group
Behavioral: Standard HIV Education & Risk Reduction — Single, individual counseling and education session. Lasting 20-30 minutes.
  Other Names: Standard HERR Counseling Session
  Arms: HIV Education & Risk Reduction Session

SUMMARY:
The MAALES Project is a community collaborative intervention designed to prevent HIV infection and transmission among African American men who have sex with both men and women. The investigators are a collaboration of researchers, community service providers and activists who are committed to developing and testing effective HIV prevention interventions that employ holistic and culturally relevant approaches. This includes recognizing the impact of forces such as racism, homophobia, heterosexism, sexism, and gender expectations on individual behavior and relationship dynamics in African American communities.

DETAILED DESCRIPTION:
HIV directly or indirectly related to male-to-male sexual intercourse is the largest contributor to HIV infection among Blacks (CDC 2002), accounting for approximately half of all US AIDS cases diagnosed among Black men and a substantial but unknown portion of cases diagnosed among Black women in 2001 (CDC 2002). The Men of African American Legacy Empowering Self (MAALES) Project is an intervention, designed to reduce HIV risk-related behaviors among African American men who have sex with men and women (MSMW) in Los Angeles.

We propose to test the efficacy of the Men of African American Legacy Empowering Self (MAALES) Project, a newly developed, novel, and culturally congruent intervention designed to reduce HIV risk-related behaviors and improve psychosocial outcomes. The MAALES intervention, which originally pilot tested with 50 men using funds from the University of California's University wide AIDS Research Program (UARP), is guided by the Theory of Reasoned Action and Planned Behavior (9; 10), the Critical Thinking and Cultural Affirmation (CTCA) Model developed by a collaborating community-based organization (11), and the Empowerment Theory (12). The small group MAALES intervention was developed through an extensive formative research process and involves six two-hour group sessions held over three weeks and lead by two ethnically matched co-facilitators. In the proposed study, we will conduct a Phase 2a test of an enhanced version of the intervention with a total of 350-400 MSMW, evenly randomized to intervention and wait listed control conditions. The enhanced intervention includes two booster sessions conducted at 1.5- and 4.5-months post conclusion of the six sessions and dialogues regarding assumptions about prospective partners' HIV serostatus. Post-intervention survey assessments will occur immediately (for psychosocial outcomes and mediators) and at three and six months post conclusion of the intervention (for all outcomes and mediators). This project will be among the first to develop and test an HIV risk-reduction intervention designed specifically for African American MSMW.

The Primary Specifics Aims are to:

1. Determine the impact of the MAALES intervention on: (a) HIV-related sexual risk behaviors and (b) sex under the influence of drugs and alcohol among African American MSMW.

   1. Hypothesis: Compared to the control condition, the MAALES Intervention condition will be more effective in decreasing episodes of unprotected anal and vaginal intercourse and number of intercourse partners at the 3- and 6-month post assessments.
   2. Hypothesis: Compared to the control condition, the MAALES Intervention condition will be more effective in decreasing the number of episodes of drug and alcohol use prior to or during sex at the 3- and 6-month post assessments.
2. Determine the impact of the MAALES intervention condition on psychosocial outcomes, including reducing HIV stigma and increasing racial/cultural pride among African American MSMW.

Hypothesis: Compared to the control condition, the MAALES Intervention condition will be more effective in decreasing HIV stigma and improving racial/cultural pride at the immediate, 3- and 6-month post assessments.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified man of African descent (black)
* 18 years of age or older
* English speaking
* Has had sex (oral, anal, mutual masturbation) with man or with a male-to-female transgender within the past 24 months.
* Has had sex (oral, anal, mutual masturbation) with a woman within the past 24 months.

Exclusion criteria:

* Participated in another HIV prevention study, in a small-group HIV prevention program or HIV prevention case management in the prior 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2007-08; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Reduced HIV-related risk sexual behaviors | 6 months
  Determine the impact of the MAALES Intervention on (a) HIV- related sexual risk behaviors and (b) sex under the influence of drugs and alcohol among African American MSMW.

SECONDARY OUTCOMES:
Internalized Homophobia | 6 months
  Examine whether reductions in internalized homophobia and gender role conflicts act as mediators of the effect of the MAALES Intervention condition on HIV risk behaviors (i.e., unprotected sexual intercourse and sex under the influence of drugs).
Psychological distress | 6 months
  Examine whether psychological distress (i.e., depression and anxiety) predicts for risky sexual behaviors and moderates the MAALES intervention condition's efficacy.
Psychosocial outcomes | 6 months
  Determine the impact of the MAALES Intervention condition on psychosocial outcomes including reducing stigma and increasing racial/cultural pride among African American MSMW.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Hawara, MPH, Ph. D, Principal Investigator — Charles Drew University; John K. Williams, MD, Principal Investigator — University of California, Los Angeles; Cleo Manago, Principal Investigator — AmASSI Health and Cultural Center; Sergio Avina, Principal Investigator — JWCH Institute, Inc.; Kevin Pickett, Principal Investigator — Palms Residential Care Facility
Locations (2):
- United States (2):
  - JWCH Institute, Inc., Los Angeles, California
  - Charles Drew University, Los Angeles, California

REFERENCES:
- [Background] Williams JK, Ramamurthi HC, Manago C, Harawa NT. Learning from successful interventions: A culturally congruent HIV risk-reduction intervention for African American men who have sex with men and women. Am J Public Health. 2009 Jun;99(6):1008-12. doi: 10.2105/AJPH.2008.140558. Epub 2009 Apr 16. PMID 19372517
- [Background] Bingham TA, Harawa NT, Williams JK. Gender role conflict among African American men who have sex with men and women: associations with mental health and sexual risk and disclosure behaviors. Am J Public Health. 2013 Jan;103(1):127-33. doi: 10.2105/AJPH.2012.300855. Epub 2012 Nov 15. PMID 23153143
- [Result] Harawa NT, Williams JK, McCuller WJ, Ramamurthi HC, Lee M, Shapiro MF, Norris KC, Cunningham WE. Efficacy of a culturally congruent HIV risk-reduction intervention for behaviorally bisexual black men: results of a randomized trial. AIDS. 2013 Jul 31;27(12):1979-88. doi: 10.1097/qad.0b013e3283617500. PMID 24180003